CLINICAL TRIAL: NCT00813384
Title: A Phase 1, First-In-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 208 in Adult Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study of AMG 208 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080895
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Oncology; Tumors; Advanced Malignancy; Advanced Solid Tumors; Oncology Patients
Keywords: Cancer; Solid Tumors; Phase 1; C-met inhibitor; Clinical Trial
MeSH Terms: conditions — Neoplasms | interventions — AMG 208

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation (Experimental): The dose escalation part of the study is aimed at determining the maximum tolerated dose (MTD), if feasible, and evaluating the safety, tolerability, pharmacokinetics and pharmacodynamics of AMG 208.
  Interventions: Drug: AMG 208
- Dose Expansion (Experimental): The dose expansion will consist of up to 30 subjects and the dose level of AMG 208 will be dependent upon emerging safety and PK data from the dose escalation part of the study.
  Interventions: Drug: AMG 208

INTERVENTIONS:
Drug: AMG 208 — AMG 208 is a small molecule inhibitor of c-Met which is a well-characterized receptor tyrosine kinase expressed on the surface of epithelial cells. C-Met receptor signaling has been shown to play a key role in the survival of cancer cells. AMG 208 inhibits both ligand-dependent and ligand-independent c-Met cellular growth regulation. Inhibition of c-Met signaling with AMG 208 provides a potential mechanism for blocking tumor growth and survival.

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of AMG 208 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Subjects must have a pathologically documented, definitively diagnosed, advanced solid tumor that is refractory to standard treatment, for which no standard therapy is available or the subject refuses standard therapy
* Measurable disease per RECIST guidelines (subjects with non-measurable, but evaluable disease are also eligible for Part 1 of the study)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Life expectancy of > 3 months, in the opinion of the investigator
* Female subjects who are post-menopausal (no menstrual period for a minimum of 12 months), or surgically sterilized. Female subjects of child bearing potential must remain abstinent or use double-barrier birth control method during the period of therapy and must be willing to use contraception 2 weeks following the last study drug administration and have a negative serum pregnancy test upon entry into this study
* Male subject is willing to use contraception upon enrollment, during the course of the study and for 12 weeks following the last study drug administration
* Willing to provide tumor samples and / or slides
* Competent to sign and date an Institutional Review Board approved informed consent form
* Hematological function, as follows:

Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Hemoglobin > 9 g/dL Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x institutional upper limit of normal (IULN)

* Renal function, as follows:

Serum creatinine < 2.0 mg/dL

* Hepatic function, as follows:

AST/ALT < 3x ULN and total bilirubin < 1.5x ULN in all subjects Alkaline phosphatase < 2.0 x ULN (if liver or bone metastases are present, ≤ 5 x ULN)

Exclusion Criteria:

* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures.
* Primary central nervous system (CNS) tumors or metastases
* History of bleeding diathesis
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication, or uncontrolled hypertension in the opinion of the investigator
* A baseline ECG QTc > 480 ms
* Active infection within 2 weeks of study enrollment (day 1)
* Significant gastrointestinal disorder(s), in the opinion of the investigator, (e.g. Crohn's disease, ulcerative colitis, extensive gastrointestinal resection) that may influence drug absorption
* Known positive test for HIV
* Known acute or chronic hepatitis B or hepatitis C infection, determined by serologic tests
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to CTCAE grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy, or investigational agent) within 28 days of study day 1 (six weeks for nitrosureas, mitomycin C, or antibody or molecular targeted agents with t1/2 > 10 days); concurrent use of hormone deprivation therapy for hormone-refractory prostate cancer or breast cancer is permitted
* Treatment with immune modulators including, but not limited to, systemic corticosteroids, cyclosporine and tacrolimus within two weeks prior to enrollment
* Therapeutic or palliative radiation therapy within 2 weeks of study day 1
* Concurrent or prior (within 7 days of study day 1) anticoagulation therapy (low-dose warfarin [≤ 2 mg/day] or low molecular weight heparins for prophylaxis against central venous catheter thrombosis or aspirin [81 mg/day] is allowed)
* Prior participation in an investigational study and/or procedure within 28 days of study day 1
* Major surgery within 30 days of study day 1
* Any co-morbid medical disorder that may increase the risk of toxicity, in the opinion of the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of AMG 208, if possible | 3.5 years
To evaluate for clinical responses associated with AMG 208 treatment in subjects (Dose Expansion) with advanced solid malignancies according to RECIST criteria | 3.5 years
To characterize the pharmacokinetic (PK) exposure of AMG 208 when administered orally to subjects with advanced solid malignancies | 3.5 years
To evaluate the safety and tolerability of AMG 208 in subjects with advanced solid malignancies | 3.5 years

SECONDARY OUTCOMES:
To evaluate for a decrease in tumor cell proliferation associated with AMG 208 treatment in subjects with advanced solid malignancies according to FLT-PET scanning | 3.5 years
To assess tumor volume changes after AMG 208 treatment by computed tomography (CT) or magnetic resonance imaging (MRI) | 3.5 years
To assess skin specimens for potential biomarkers | 3.5 years
To determine whether c-Met expression, mutation, or amplification in tumor specimens correlates with a response to AMG 208 | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Beverly Hills, California
  - Research Site, St Louis, Missouri
  - Research Site, Houston, Texas

REFERENCES:
- [Derived] Hong DS, Rosen P, Lockhart AC, Fu S, Janku F, Kurzrock R, Khan R, Amore B, Caudillo I, Deng H, Hwang YC, Loberg R, Ngarmchamnanrith G, Beaupre DM, Lee P. A first-in-human study of AMG 208, an oral MET inhibitor, in adult patients with advanced solid tumors. Oncotarget. 2015 Jul 30;6(21):18693-706. doi: 10.18632/oncotarget.4472. PMID 26155941
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com